CLINICAL TRIAL: NCT06595862
Title: Development and Evaluation of an Avatar-guided Mobile Health Intervention for Emerging Adults With Alcohol Misuse and Suicidality
Brief Title: Open Pilot Trial Evaluating an Avatar-Guided Intervention for Emerging Adults With Alcohol Use Problems and Suicide Risk
Acronym: EA-Avatar
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Lourah Kelly, Assistant Professor, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 001128; R00AA029154 (NIH)
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Binge Drinking; Suicidal Ideation
Keywords: alcohol; suicidal thoughts; open pilot trial
MeSH Terms: conditions — Binge Drinking; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: This is a single group open pilot trial, in order to test the usability of the EA-Avatar digital intervention and feasibility of the research protocols of the EA-Avatar intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EA-Avatar (Experimental): The avatar-guided digital intervention includes monitoring of alcohol use and common triggers suicidal thoughts, skills to manage alcohol use and suicidal thoughts, resources on how to access outpatient care and crisis hotlines for suicidal thoughts, and achievements for milestones. In addition, text messages provide reminders to access the avatar platform to learn or practice skills and provide encouragement. EA-Avatar is given in addition to emergency department care as usual.
  Interventions: Behavioral: EA-Avatar

INTERVENTIONS:
Behavioral: EA-Avatar — The avatar-guided digital intervention includes monitoring of alcohol use and common triggers suicidal thoughts, skills to manage alcohol use and suicidal thoughts, resources on how to access outpatient care and crisis hotlines for suicidal thoughts, and achievements for milestones. In addition, text messages provide reminders to access the avatar platform to learn or practice skills and provide encouragement.

SUMMARY:
This study is an open pilot usability trial to test the 1) usability of a newly developed mobile health intervention to help manage suicidal ideation and alcohol use problems and 2) feasibility of research protocols with emerging adults (18-29 year-olds) who present to the emergency department.

DETAILED DESCRIPTION:
This study is an open pilot usability trial with emerging adults presenting to the emergency department with binge drinking and suicidal thoughts. The main study aims are to test the usability of a newly developed avatar-guided mobile health intervention and feasibility of 28 days of daily assessments and four follow-ups at 4-, 8-, and 12-weeks after discharge.

Ten emerging adults aged 18-29 years old will be recruited from the emergency department who have suicidal ideation and alcohol use problems. Exclusion criteria are conditions that would preclude research participation (e.g., cognitive disabilities, in police custody; at imminent risk of harming oneself in the emergency department).

All ten participants will be given access to a newly designed avatar-guided digital intervention and text message intervention (EA-Avatar) for 12 weeks in addition to usual emergency department care. Participants will complete measures of alcohol use, suicidal ideation, and alcohol-related cognitions and experiences, as well as service utilization. They will also complete a scale of usability of the avatar intervention and qualitative interviews of the intervention and research protocols.

Based on participant qualitative interviews, a scale of usability of the digital intervention, feedback surveys, recruitment and retention in the study, participant completion of daily diary and ecological assessment surveys, and analysis of mobile intervention usage data, the intervention will be revised, before testing in a larger randomized controlled feasibility trial.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-29 years old
* Past month binge drinking OR score of 6 or greater on the Alcohol Use Disorder Identification Test
* Past month active suicidal ideation per clinical chart and confirmed via self-report
* Have a personal smartphone device with internet access
* Speak, read, and understand English

Exclusion Criteria:

* Severe cognitive delay, active psychosis, or heavy intoxication that would interfere with understanding the study
* Imminent safety risk requiring a 1:1 observation
* In police custody during emergency department visit
* Unwilling or not interested in using an avatar-directed intervention in addition to their usual emergency department care

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Usability of the EA-Avatar digital intervention, defined by ratings on the System Usability Scale | 12 weeks
  If any System Usability Items are less than 3.5 out of 5, those aspects of the digital intervention will be revised in the beta version.
Feasibility of research protocols, defined as follow-up retention | 12 weeks
  Feasibility will be supported by retention of research participants in at least 80% at each of the four assessments
Feasibility of research protocols, defined as adherence to the ecological momentary assessment/daily diary protocol | 12 weeks
  Feasibility will be supported by at least 75% of total EMA and daily diary surveys across 28 days

SECONDARY OUTCOMES:
Acceptability of EA-Avatar as rated on participant feedback surveys | 12 weeks
  Feedback on the alpha version of EA-Avatar measured via a feedback survey with items rated on a 4-point likert scale from strongly disagree to strongly agree, which assesses opinions about avatar appearance and customizations, the helpfulness of skills, and helpfulness of features of the platform

CONTACTS AND LOCATIONS:
Overall Officials: Lourah M. Kelly, Principal Investigator — UMass Worcester (UMass Chan Medical School)
Locations (2):
- United States (2):
  - UMass Memorial Health - Marlborough Hospital, Marlborough, Massachusetts
  - UMass Memorial, University Campus, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with per reasonable request to the PI, after the final report and data is published in a peer-reviewed scientific journal.
Supporting Information: Study Protocol, ICF
Time Frame: 6 months after the last participant completes the study (completes their 12 week follow-up), data will be analyzed and submitted for publication in a peer-reviewed scientific journal.
Access Criteria: After publication of main and secondary outcomes in a peer-reviewed journal, de-identified data will be available upon reasonable request to the PI.